CLINICAL TRIAL: NCT06500195
Title: Cobb Angle Comparison of Hybrid Construct Versus Pedicle Screw-only System for the Treatment of Lenke 1 Adolescent Idiopathic Scoliosis
Brief Title: Hybrid Construct Versus Pedicle Screw-only System for the Treatment Scoliosis
Status: Completed | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Sponsor
Other Study IDs: KB.006.112.2023
Record Dates: First submitted 2024-07-02; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Scoliosis Idiopathic; Dysplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SCREWS: The SCREWS group of patients operated on with the use of only transpedicular screws.
- HYBRID: The HYBRID group of patients whose corrections were performed using the hybrid instrumentation system (screws and bands).
  Interventions: Procedure: implantation of the hybrid instrumentation system

INTERVENTIONS:
Procedure: implantation of the hybrid instrumentation system — Surgery corrections were performed using the hybrid instrumentation system (screws and bands).
  Groups: HYBRID

SUMMARY:
The placement of pedicular screws in spinal surgery has become the gold standard for scoliosis treatment. However, the use of sublaminar bands (SBs) on the apex of the curvature in idiopathic scoliosis (AIS) lowers the risk of neurological complications related to incorrect implementation of transpedicular screws into dysplastic pedicles without a cancellous channel. The latest research does not define a set of anatomical guidelines for applying SBs, nor does it use a dedicated classification system related to the structure of pedicles. The aim of this study was to assess the safety of the method and the correction attained through hypoplastic/aplastic pedicles when applying a hybrid instrumentation system to patients suffering from AIS Lenke type 1. Methods: Twenty patients were involved in a prospective, single-center, non-randomized case series study. The patients were assigned to the group "SCREWS" or "HYBRID" where SBs were used.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is a three-dimensional deformation of the spine. The goal of the treatment is to achieve a reduction in deformity, restoring proper alignment and the best possible function of the spine. Pedicular screw placement in spinal surgery has become the gold standard for scoliosis reduction techniques in the last 30 years [6]. The screw-only systems are relatively safe, as various authors have proven. However, if implemented incorrectly, the screws increase the risk of damage to nervous or vascular structures and internal organs. The latest research does not define a set of anatomical guidelines for applying SBs, nor does it use a dedicated classification system related to the structure of pedicles. The aim of this study was to assess the safety of the method and the correction attained through hypoplastic/aplastic pedicles when applying a hybrid instrumentation system to patients suffering from AIS Lenke type 1. Methods: Twenty patients were involved in a prospective, single-center, non-randomized case series study. The patients were assigned to the group "SCREWS" or "HYBRID" where SBs were used. The inclusion criteria were this being the patients' first scoliosis operation due to AIS (Lenke type 1) and age under 18 years. The primary measured outcome involved correction efficacy, defined as the Cobb score baseline to endpoint change.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic scoliosis (AIS)
* Lenke type 1

Exclusion Criteria:

* AIS other than Lenke type 1 (neurogenic, congenial, or syndromic curvatures)
* abnormalities in the structure of the central nervous system in the MRI image
* advanced chronic respiratory or circulatory failure
* emergency surgery
* reoperation

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who qualified for scoliosis surgery in this center underwent X-ray imaging (AP, lateral, lateral bending view), computed tomography, and magnetic resonance imaging. Patients with a Cobb angle greater than 45 degrees (or 40 degrees in highly progressive cases) were considered eligible for the study. Based on the computed tomography assessment that was performed prior to the surgery, patients were assigned to one of two groups depending on the pedicle type on the apex of the thoracic curvature according to Watanabe pedicle's classification.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
correction efficacy | at the 3rd day after the surgery procedure
  defined as the Cobb score baseline to endpoint change (Cobb angle change in the operated spine segment in % at endpoint: X-ray imaging was performed (AP and lateral)

SECONDARY OUTCOMES:
length of surgery procedure | procedure (from skin incision to skin suture)
  duration of the hospitalization measured in minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Pomeranian Medical University, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: Undecided
after personal request